CLINICAL TRIAL: NCT00802906
Title: Prospective Study on the Efficacy of 1.5mg Bevacizumab Versus Selective Subthreshold Micropulslaser in Central Serous Chorioretinopathy
Brief Title: Bevacizumab Versus Micropulse in Central Serous Chorioretinopathy (CSC)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Michael Koss, PI, Johann Wolfgang Goethe University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MK-RCS-2008
Record Dates: First submitted 2008-12-04; First posted 2008-12-05 (Estimated); Last update posted 2012-09-27 (Estimated); Status verified 2012-09

CONDITIONS: Central Serous Chorioretinopathy
Keywords: micropulselaserphotocoagulation; bevacizumab; CSC
MeSH Terms: conditions — Central Serous Chorioretinopathy | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): 1.5 mg bevacizumab single injection and on demand if leakage is persistent or recurs
  Interventions: Device: subthreshold micropulselaser; Drug: bevacizumab
- 2 (Active Comparator): initial selective subthreshold micropulselasercoagulation and on demand if leakage is persistent or recurs
  Interventions: Device: subthreshold micropulselaser
- 3 (No Intervention): control

INTERVENTIONS:
Device: subthreshold micropulselaser — on demand if leakage is persistent or recurs after initial treatment
  Arms: 1; 2
Drug: bevacizumab — 1.5 mg initial intravitreal injection
  Arms: 1

SUMMARY:
The purpose of this study is to evaluate the clinical efficacy of an initial subthreshold retinal micropulselasercoagulation versus a single intravitreal 1.5mg bevacizumab injection in central serous choriretinopathy, as the micropulse will selectively treat the damaged RPE to induce reproliferation of healthy RPE cells, whereas the intravitreal injection should non-selectively stop the RPE leakage.

DETAILED DESCRIPTION:
To evaluate the clinical efficacy of an initial subthreshold retinal micropulselasercoagulation in twelve eyey per group versus a single intravitreal 1.5mg bevacizumab injection in central serous choriretinopathy, as the micropulse will selectively treat the damaged RPE to induce reproliferation of healthy RPE cells. BCVA in EDTRS score, OCT, and leakage in FLA, static perimetry of both groups will be correlated to a control group without treatment over 10 months.

ELIGIBILITY:
Inclusion criteria:

* CSC of >4 months duration

Exclusion Criteria:

* History of macular or chorioretinal inflammation
* Lens / corneal opacities

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-05; Primary Completion 2010-11 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
BCVA in EDTRS values | 24 months

SECONDARY OUTCOMES:
OCT, leakage in FA, defects in satic perimetry | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Koss, MD, Principal Investigator — ZAU Department of Vitreoretinal surgery
Locations (1):
- ZAU Department of VR surgery, Frankfurt am Main, Hesse, Germany

REFERENCES:
- [Derived] Koss MJ, Beger I, Koch FH. Subthreshold diode laser micropulse photocoagulation versus intravitreal injections of bevacizumab in the treatment of central serous chorioretinopathy. Eye (Lond). 2012 Feb;26(2):307-14. doi: 10.1038/eye.2011.282. Epub 2011 Nov 11. PMID 22079961